CLINICAL TRIAL: NCT04323917
Title: Detection of High Expression Levels of EMT-Transcription Factor mRNAs in Patients With Pancreatic Cancer and Their Diagnostic Potential
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: EMT PC 1.1
Record Dates: First submitted 2019-12-20; First posted 2020-03-27 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Cancer
Keywords: Epithelial to Mesenchymal Transition; EMT; PC; mRNA; EMT-TF; Diagnosis; Biomarkers; Liquid biopsy
MeSH Terms: conditions — Pancreatic Neoplasms; Disease | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — mRNA from whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Subjects affected by Pancreatic carcinoma (PC) confirmed by tissue biopsy
  Interventions: Diagnostic Test: Liquid biopsy
- Controls: Healthy Subject enrolled following colon cancer screening via colonoscopy
  Interventions: Diagnostic Test: Liquid biopsy

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — Detection and quantification of EMT-transcription factor mRNA levels in blood

SUMMARY:
The present study is aimed at detecting and measuring mRNA levels of genes involved in epithelial to mesenchymal transition (EMT) in biological samples, i.e. in peripheral blood samples of pancreatic cancer (PC) patients and healthy controls, to determine the presence of disease, its progression and risk of recurrence.

DETAILED DESCRIPTION:
The investigators first provided evidence that human pancreatic cancer (PC) cells can undergo EMT during local invasion, and that EMT transcription factors (i.e.Twist family basic helix-loop-helix transcription factor 1 (TWIST1)) are increased in the blood of PC patients. In addressing the relevance of EMT in the metastatic process, the prognostic role of M-like cancer cells entering into the circulation remains to be determined.

Currently, the notion that cancer disseminates via the circulation led to increased attention on the identification of circulating tumor cells (CTCs) in blood samples ("liquid biopsy"; LB), so far exclusively based upon epithelial (E) markers. However, an un-biased evaluation of CTCs, providing meaningful information for cancer diagnosis up to therapy, cannot exclude cells with M features. LB data show that circulating TWIST1, zinc finger E-box binding homeobox 2 (ZEB2) and E-Cadherin (CDH1) messenger ribonucleic acids (mRNA) are significantly and steadily increased in the blood of PC patients.These findings indicate that high levels of EMT players in the circulation efficiently discriminate PC patients, irrespectively of tumor resectability.

The present study is aimed at detecting and measuring mRNA levels of genes involved in epithelial to mesenchymal transition in biological samples, i.e. in peripheral blood samples of tumor patients, to determine the presence of disease, its progression and risk of recurrence.

Aim of the study is to depict the molecular profile of EMT-Transcription factor (EMT-TFs) variations in the blood of patients with early, intermediate or advanced PC, with respect to disease progression and delivered treatments.

Primary endpoint: to determ the stage, the remission or the progression of a pancreatic cancer in a pancreatic cancer affected subjects. This end-point comprising the step of assaying a biological sample from said subject for the presence of a panel of mRNAs encoding for transcription factors involved in epithelial to mesenchymal transition.

Secondary endpoint: to identify biomarkers suitable for the selection of patients amenable of responsiveness to medical and surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females over 18 years of age capable of providing informed consent.
2. Pancreatic carcinoma confirmed by tissue biopsy or colon mass, clinically consistent with cancer and eventually confirmed by pathology.
3. Subject were enrolled following colon cancer screening via colonoscopy

Exclusion Criteria:

1. Patients under the age of 18 years or over the age of 80 years.
2. Patients with personal history of cancer, identification of large polyp or adenomatous pathology on previous or subsequent colonoscopy
3. Patient with history of abdominal surgery within the past four months
4. Patients unwilling to or unable to give informed consent.
5. Patients with acute inflammatory diseases or under any emergency condition.
6. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective pathological and molecular study of screening for pancreatic cancer. The main objectives of the trial are:
  1. To develop a specific and reproducible assay for the detection pancreatic cancer based on blood RNA and to amplify cancer specific molecular markers using qPCR.
  2. To correlate the presence of molecular markers in the samples with the presence of pancreatic cancer or pre-cancerous lesions.
  3. To add additional biomarkers to the study panel of biomarkers. presence of colon cancer or pre-cancerous lesions. To add additional biomarkers to the study panel of biomarkers.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Assessments of diagnosis of PC by EMT-TF mRNA levels in blood | Analysis at day 0: at diagnosis or before surgery for PC patients; before colonoscopy in controls
  To determine the stage, the remission or the progression of a pancreatic cancer in a pancreatic cancer affected subject not administered with an appropriate antitumor treatment (e.g., neo-adjuvant therapy) comprising the step of assaying a biological sample from said subject for the presence of a panel of mRNAs encoding for transcription factors involved in epithelial to mesenchymal transition.

SECONDARY OUTCOMES:
Prediction of prognosis of PC by EMT-TF mRNA levels in blood | Analysis at least: 7-15 days from surgery (T1), 30 days (T2) from surgery, 6 months (T3) from surgery, 1 year (T4) from surgery
  To identify biomarkers suitable for the selection of PC patients amenable of responsiveness to medical and surgical treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico humanitas, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Data patent covered. No. Patent: EP13197367.9 - December 16, 2013

REFERENCES:
- [Background] Celesti G, Di Caro G, Bianchi P, Grizzi F, Basso G, Marchesi F, Doni A, Marra G, Roncalli M, Mantovani A, Malesci A, Laghi L. Presence of Twist1-positive neoplastic cells in the stroma of chromosome-unstable colorectal tumors. Gastroenterology. 2013 Sep;145(3):647-57.e15. doi: 10.1053/j.gastro.2013.05.011. Epub 2013 May 15. PMID 23684708